CLINICAL TRIAL: NCT03472326
Title: A Phase 2 Study to Evaluate the Efficacy of GS-9131 Functional Monotherapy in HIV-1-Infected Adults Failing a Nucleos(t)Ide Reverse Transcriptase Inhibitor-Containing Regimen With Nucleos(t)Ide Reverse Transcriptase Inhibitor Resistant Virus
Brief Title: Study to Evaluate the Efficacy of GS-9131 Functional Monotherapy in Human Immunodeficiency Virus (HIV)-1-Infected Adults Failing a Nucleos(t)Ide Reverse Transcriptase Inhibitor-Containing Regimen With Nucleos(t)Ide Reverse Transcriptase Inhibitor Resistant Virus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: GS-9131 did not meet the targeted antiviral response
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-442-4148
Record Dates: First submitted 2018-03-08; First posted 2018-03-21 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — GS-9131; imidazole mustard; tenofovir alafenamide; Darunavir; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Sentinel Cohort 1: GS-9131 60 mg (Experimental): Treatment experienced participants will receive GS-9131 60 mg in addition to their current failing ARV regimen for a period of 10 days.
  Interventions: Drug: GS-9131; Drug: ARV regimen
- Part 1 Sentinel Cohort 2: GS-9131 180 mg (Experimental): Treatment experienced participants will receive GS-9131 180 mg in addition to their current failing ARV regimen for a period of 14 days.
  Interventions: Drug: GS-9131; Drug: ARV regimen
- Part 1: Randomized Cohort (Experimental): Participants will be randomized in 1:1:1:1 so as to receive GS-9131 in 3 active dose levels up to a maximum of 180 mg or Placebo to match GS-9131 in addition to their current failing ARV regimen for a period of 14 days in Part 1.
  Interventions: Drug: GS-9131; Drug: ARV regimen
- Part 2 Sentinel Cohort 1: GS-9131 + BIC + DRV + RTV (Experimental): Participants who complete dosing in Sentinel Cohort 1 of Part 1 and show a reduction in plasma HIV RNA > 0.5 log10 from their pre-GS-9131 baseline value at Day 11 and discontinue their current failing regimen will receive an optimized regimen consisting of GS-9131 60 mg + bictegravir (BIC) 30 mg + darunavir (DRV) 800 mg + ritonavir (RTV) 100 mg for a period of 24 weeks. After Week 24, participants will be given the option to participate in an open label extension and receive GS-9131 60 mg + BIC 75 mg + tenofovir alafenamide (TAF) 25 mg, for an additional 24 weeks or until Gilead Sciences elects to discontinue the study drug in that country, whichever occurs first.
  Interventions: Drug: GS-9131; Drug: BIC; Drug: DRV; Drug: RTV
- Part 2 Sentinel Cohort 2: GS-9131 + BIC + TAF (Experimental): Participants who complete dosing in Sentinel Cohort 2 of Part 1 and show a reduction in plasma HIV RNA > 0.5 log10 from their pre-GS-9131 baseline value at Day 15 and discontinue their current failing regimen will receive an optimized regimen consisting of GS-9131 180 mg + BIC 75 mg + TAF 25 mg, for a period of 24 weeks. After Week 24, participants will be given the option to participate in an open label extension and receive GS-9131 180 mg + BIC 75 mg + TAF 25 mg, for an additional 24 weeks or until Gilead Sciences elects to discontinue the study drug in that country, whichever occurs first.
  Interventions: Drug: GS-9131; Drug: BIC; Drug: TAF

INTERVENTIONS:
Drug: GS-9131 — Tablet(s) administered orally once daily
Drug: BIC — Tablet(s) administered orally once daily
  Arms: Part 2 Sentinel Cohort 1: GS-9131 + BIC + DRV + RTV; Part 2 Sentinel Cohort 2: GS-9131 + BIC + TAF
Drug: TAF — Tablet(s) administered orally once daily
  Other Names: Vemlidy®
  Arms: Part 2 Sentinel Cohort 2: GS-9131 + BIC + TAF
Drug: ARV regimen — ARV regimen may consist of the ARV agents containing nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) and non-nucleoside reverse transcriptase inhibitor (NNRTI)
  Arms: Part 1 Sentinel Cohort 1: GS-9131 60 mg; Part 1 Sentinel Cohort 2: GS-9131 180 mg; Part 1: Randomized Cohort
Drug: DRV — Tablet(s) administered orally once daily
  Other Names: Prezista®
  Arms: Part 2 Sentinel Cohort 1: GS-9131 + BIC + DRV + RTV
Drug: RTV — Tablet(s) administered orally once daily
  Other Names: Norvir®
  Arms: Part 2 Sentinel Cohort 1: GS-9131 + BIC + DRV + RTV

SUMMARY:
The primary objective of this study is to evaluate the short-term antiviral potency of GS-9131 functional monotherapy compared to placebo-to-match (PTM) GS-9131, each administered once daily with the existing failing antiretroviral (ARV) regimen as demonstrated by the proportion of participants achieving human immunodeficiency virus ribonucleic acid (HIV-1 RNA) > 0.5 log10 decreases from baseline after up to 14 days of therapy in HIV-1 positive, ARV treatment experienced adult participants with nucleos(t)ide resistant virus.

This is a two-part study. Part 1 consists of three cohorts: 2 Sentinel Cohorts and 1 Randomized Cohort. Eligible participants from Part 1 will proceed to Part 2 followed by an optional open-label extension.

ELIGIBILITY:
Key Inclusion Criteria:

* Plasma HIV-1 RNA ≥ 500 copies/mL at screening Visit
* Currently taking a failing ARV regimen that contains 2 NRTIs and a NNRTI
* No prior or current ARV regimens containing integrase inhibitor (INSTI) or protease inhibitor (PI)
* Screening genotype must show at least the protocol defined resistance mutation profile

Key Exclusion Criteria:

* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Day 1
* Participation in any other clinical trial, including observational studies, without prior approval from the sponsor is prohibited while participating in this trial
* Use of an investigational drug other than the study drug
* Individuals with chronic hepatitis B virus (HBV) infection are not permitted to participate
* Active tuberculosis infection

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (2):
- Joint Clinical Research Centre, Kampala, Uganda
- Joint Research Ethics Committee for the University of Zimbabwe College of Health Sciences and Parirenyatwa Group of Hospitals, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Uganda and Zimbawe. The first participant was screened on 03 April 2018. The last study visit occurred on 09 December 2019.
Pre-assignment Details: 88 participants were screened. The study was conducted in 2 parts. The Part 1 consisted of 3 cohorts- 2 Sentinel Cohorts and 1 Randomized Cohort and Part 2 consisted of 2 Sentinel Cohorts only. The Randomized Cohort in Part 1 was not initiated. The study was terminated because a majority of Sentinel Cohort 2 (Part 1) participants did not meet primary endpoint of human immunodeficiency virus ribonucleic acid (HIV-1 RNA) > 0.5 log10 decrease from baseline in through up to 14 days of therapy.
Groups:
- Part 1 Sentinel Cohort 1: GS-9131 60 mg: Participants received GS-9131 60 mg tablets orally once daily in addition to their current failing antiretroviral (ARV) regimen for a period of 10 days.
- Part 1 Sentinel Cohort 2: GS-9131 180 mg: Participants received GS-9131 180 mg tablets orally once daily in addition to their current failing ARV regimen for a period of 14 days.
- Part 2 Sentinel Cohort 1: GS-9131 + BIC + DRV + RTV: Participants who completed dosing in Sentinel Cohort 1 and showed a reduction in plasma HIV RNA > 0.5 log10 from their pre-GS-9131 baseline value at Day 11 and discontinued their current failing regimen received an optimized regimen consisting of GS-9131 60 mg tablets + bictegravir (BIC) 30 mg tablets + darunavir (DRV) 800 mg tablets + ritonavir (RTV) 100 mg tablets, orally once daily for a period of 24 weeks. After Week 24, participants had the option to participate in an open label extension and receive GS-9131 60 mg tablets + BIC 75 mg tablets + tenofovir alafenamide (TAF) 25 mg tablets, orally once daily for an additional 24 weeks or until Gilead Sciences elects to discontinue the study drug in that country, whichever occurred first.
- Part 2 Sentinel Cohort 2: GS-9131 + BIC + TAF: Participants who completed dosing in Sentinel Cohort 2 and showed a reduction in plasma HIV RNA > 0.5 log10 from their pre-GS-9131 baseline value at Day 15 and discontinued their current failing regimen received an optimized regimen consisting of GS-9131 180 mg tablets + BIC 75 mg tablets + TAF 25 mg tablets, orally once daily for a period of 24 weeks. After Week 24, participants had the option to participate in an open label extension and receive GS-9131 180 mg tablets + BIC 75 mg tablets + TAF 25 mg tablets, orally once daily for an additional 24 weeks or until Gilead Sciences elects to discontinue the study drug in that country, whichever occurred first.
Period: Part 1: GS-9131 Functional Monotherapy
Arm/Group | Part 1 Sentinel Cohort 1: GS-9131 60 mg | Part 1 Sentinel Cohort 2: GS-9131 180 mg | Part 2 Sentinel Cohort 1: GS-9131 + BIC + DRV + RTV | Part 2 Sentinel Cohort 2: GS-9131 + BIC + TAF
Started | 11 | 10 | 0 | 0
Completed | 11 | 10 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2: Combination Therapy
Arm/Group | Part 1 Sentinel Cohort 1: GS-9131 60 mg | Part 1 Sentinel Cohort 2: GS-9131 180 mg | Part 2 Sentinel Cohort 1: GS-9131 + BIC + DRV + RTV | Part 2 Sentinel Cohort 2: GS-9131 + BIC + TAF
Started | 0 | 0 | 1 (Of the participants who completed Part 1, only 1 participant entered in Part 2.) | 3 (Of the participants who completed Part 1, only 3 participants entered in Part 2.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 3
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study medication.
Groups:
- Sentinel Cohort 1: GS-9131 60 mg: Participants in Sentinel Cohort 1 received GS-9131 60 mg tablets orally once daily in addition to their current failing ARV regimen for a period of 10 days in Part 1.
- Sentinel Cohort 2: GS-9131 180 mg: Participants in Sentinel Cohort 2 received GS-9131 180 mg tablets orally once daily in addition to their current failing ARV regimen for a period of 14 days in Part 1.
- Total: Total of all reporting groups
Arm/Group | Sentinel Cohort 1: GS-9131 60 mg | Sentinel Cohort 2: GS-9131 180 mg | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (10.7) | 37 (6.6) | 38 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 11 | 5 | 16
  Zimbabwe | 0 | 5 | 5
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.77 (0.703) | 4.46 (0.584) | 4.62 (0.652)
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 0 | 0 | 0
  ≥ 50 copies/mL | 11 | 10 | 21
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 172 (164.1) | 289 (140.4) | 228 (161.0)

OUTCOME MEASURES:

1. Primary Outcome: Part 1 Randomized Cohort: Percentage of Participants With Plasma HIV-1 RNA Decreases From Baseline Exceeding 0.5 log10 at Day 15
Description: The criteria for analyzing percentage of participants with plasma HIV-1 RNA > 0.5 log10 decrease from baseline in randomized cohort was at least 50% of the participants should achieve HIV-1 RNA > 0.5 log10 decrease from baseline in the Part 1 sentinel cohort 2.
Time Frame: Day 15
Population: Data was not analyzed as ≥ 50% participants did not achieve HIV-1 RNA > 0.5 log10 decrease from baseline in Part 1 sentinel cohort 2.
Groups:
- Part 1: Randomized Cohort: Participants were randomized in 1:1:1:1 so as to receive GS-9131 tablets orally once daily in 3 active dose levels up to a maximum of 180 mg or Placebo to match GS-9131 tablets orally once daily in addition to their current failing ARV regimen for a period of 14 days in Part 1.
Arm/Group | Part 1: Randomized Cohort
Number analyzed (Participants) | 0

2. Secondary Outcome: Part 1 Sentinel Cohort 1: Change From Baseline in Plasma log10 HIV-1 RNA at Day 11
Time Frame: Baseline, Day 11
Population: The Safety Analysis Set included all participants who took at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Sentinel Cohort 1: GS-9131 60 mg
Number analyzed (Participants) | 11
log10 copies/mL | -0.13 (0.268)

3. Secondary Outcome: Part 1 Sentinel Cohort 2: Change From Baseline in Plasma log10 HIV-1 RNA at Day 15
Time Frame: Baseline, Day 15
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Sentinel Cohort 2: GS-9131 180 mg
Number analyzed (Participants) | 8
log10 copies/mL | -0.29 (0.207)

4. Secondary Outcome: Part 1 Randomized Cohort: Change From Baseline in Plasma log10 HIV-1 RNA at Day 15
Time Frame: Baseline, Day 15
Population: Data was not reported as the Randomized Cohort in Part 1 was not initiated as the study was terminated early because a majority of Sentinel Cohort 2 participants did not meet primary endpoint of HIV-1 RNA > 0.5 log10 decrease from baseline in through up to 14 days of therapy.
Arm/Group | Part 1: Randomized Cohort
Number analyzed (Participants) | 0

5. Secondary Outcome: Part 2: Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL as Defined by the FDA Snapshot Analysis at Week 24
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Data were collected for only 1 participant, and due to participant confidentiality data is not being reported.
Groups:
- Part 2: GS-9131 + BIC + DRV + RTV: Participants who completed dosing in Sentinel Cohort 1 and showed a reduction in plasma HIV RNA > 0.5 log10 from their pre-GS-9131 baseline value at Day 11 and discontinued their current failing regimen received an optimized regimen consisting of GS-9131 60 mg tablets + BIC 30 mg tablets + DRV 800 mg tablets + RTV 100 mg tablets, orally once daily for a period of 24 weeks. After Week 24, participants will be given the option to participate in an open label extension and receive GS-9131 60 mg tablets + BIC 75 mg tablets + TAF 25 mg tablets, orally once daily for an additional 24 weeks or until Gilead Sciences elects to discontinue the study drug in that country, whichever occurred first.
- Part 2: GS-9131 + BIC + TAF: Participants who completed dosing in Sentinel Cohort 2 and showed a reduction in plasma HIV RNA > 0.5 log10 from their pre-GS-9131 baseline value at Day 15 and discontinued their current failing regimen received an optimized regimen consisting of GS-9131 180 mg tablets + BIC 75 mg tablets + TAF 25 mg tablets, orally once daily for a period of 24 weeks. After Week 24, participants will be given the option to participate in an open label extension and receive GS-9131 180 mg tablets + BIC 75 mg tablets + TAF 25 mg tablets, orally once daily for an additional 24 weeks or until Gilead Sciences elects to discontinue the study drug in that country, whichever occurred first.
Arm/Group | Part 2: GS-9131 + BIC + DRV + RTV | Part 2: GS-9131 + BIC + TAF
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Part 2: Change From Baseline in Plasma log10 HIV-1 RNA at Week 24
Time Frame: Baseline, Week 24
Population: Data were collected for only 1 participant, and due to participant confidentiality data is not being reported.
Arm/Group | Part 2: GS-9131 + BIC + DRV + RTV | Part 2: GS-9131 + BIC + TAF
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Part 2: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline, Week 24
Population: Data were collected for only 1 participant, and due to participant confidentiality data is not being reported.
Arm/Group | Part 2: GS-9131 + BIC + DRV + RTV | Part 2: GS-9131 + BIC + TAF
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Part 2: Number of Participants With Treatment Emergent Nucleos(t)Ide Reverse Transcriptase Inhibitor (NRTI) Mutations at the Time of Virologic Failure
Description: Treatment emergent virological failure was defined as an event with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of the study drug. Virologic failure was defined as virologic rebound or as suboptimal virologic response in relation to pre-GS-9131 baseline plasma HIV-1 RNA levels. Virological rebound was defined as if participant at any visit after achieving HIV-1 RNA < 50 copies/mL, a rebound in HIV-1 RNA ≥ 50 copies/mL, or a >1 log10 increase in HIV-1 RNA from the nadir which was subsequently confirmed at the following scheduled or unscheduled visit. Suboptimal virologic response was defined as plasma HIV-1 RNA ≥ 200 copies/mL and reduction in HIV-1 RNA ≤ 1 log10 from pre-GS-9131 baseline at the Week 8 visit with confirmation at the next scheduled or unscheduled visit.
Time Frame: From first dose up to Week 24
Population: Due to early study termination, data were not collected as none of the participants qualified for resistance testing after Week 8.
Arm/Group | Part 2: GS-9131 + BIC + DRV + RTV | Part 2: GS-9131 + BIC + TAF
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Part 2: Number of Participants With Treatment Emergent Protease Inhibitor (PI) Mutations at the Time of Virologic Failure
Description: as for outcome 8
Time Frame: From first dose up to Week 24
Population: as for outcome 8
Arm/Group | Part 2: GS-9131 + BIC + DRV + RTV | Part 2: GS-9131 + BIC + TAF
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Part 2: Number of Participants With Treatment Emergent Integrase Strand Transfer Inhibitor (INSTI) Mutations at the Time of Virologic Failure
Description: as for outcome 8
Time Frame: From first dose up to Week 24
Population: as for outcome 8
Arm/Group | Part 2: GS-9131 + BIC + DRV + RTV | Part 2: GS-9131 + BIC + TAF
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose date up to 30 days after last study drug for Part 1 (Maximum: 44 days)
Description: The Safety Analysis Set included all participants (in Sentinal Cohorts 1 and 2 in part 1) who took at least 1 dose of study medication. Due to the early discontinuation of the study, safety analyses were performed for Sentinel Cohorts in Part 1 only. In Part 2, Data were collected for only 1 participant, and due to participant confidentiality data is not being reported.
Groups:
- Part 1 Setinel Cohort 1: GS-9131 60 mg: Participants in Sentinel Cohort 1 received GS-9131 60 mg tablets orally once daily in addition to their current failing ARV regimen for a period of 10 days in Part 1.
- Part 1 Sentinel Cohort 2: GS-9131 180 mg: Participants in Sentinel Cohort 2 received GS-9131 180 mg tablets orally once daily in addition to their current failing ARV regimen for a period of 14 days in Part 1.
Arm/Group | Part 1 Setinel Cohort 1: GS-9131 60 mg | Part 1 Sentinel Cohort 2: GS-9131 180 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 5/11 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Setinel Cohort 1: GS-9131 60 mg (N=11) | Part 1 Sentinel Cohort 2: GS-9131 180 mg (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Malaise (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Amylase increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 1 | 2
Hypersomnia (Nervous system disorders) | 0 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Pica (Psychiatric disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated because a majority of Sentinel Cohort 2 participants did not meet primary endpoint of HIV-1 RNA > 0.5 log10 decrease from baseline through up to 14 days of therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT03472326/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT03472326/SAP_001.pdf